CLINICAL TRIAL: NCT06823466
Title: Advancing Knowledge in Ischemic Stroke Patients on Oral Anticoagulants - The ASPERA International Registry
Brief Title: Advancing Knowledge in Ischemic Stroke Patients on Oral Anticoagulants
Acronym: ASPERA
Status: Recruiting | Type: Observational
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Simona Sacco, Professor, University of L'Aquila
Other Study IDs: 2696 - 22/07/2024
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Oral Anticoagulation; Atrial Fibrillation (AF); Outcome Assessment; Clinical Presentations
Keywords: Ischemic stroke; Oral anticoagulation; Atrial fibrillation; Direct oral anticoagulants; Vitamin k antagonists; Outcomes; Prognosis; Clinical characteristics; Secondary prevention
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASPERA-R: Retrospectively enrolled schemic stroke patients on oral anticoagulants at the time of the index stroke followed up at hospital discharge and 90 days post-stroke
- ASPERA-P: Prospectively enrolled ischemic stroke patients on oral anticoagulants at the time of the index stroke followed up at 90 days, 1 year and 5 years post-stroke

SUMMARY:
The Advancing knowledge in ischemic Stroke PatiEnts on oRal Anticoagulants (ASPERA) study aims to investigate characteristics of ischemic stroke cases occurring in patients on oral anticoagulation for atrial fibrillation (AF) or other cardioembolic arrhythmias and to characterize short and long-term outcomes associated with different secondary prevention strategies to prevent stroke recurrences. The ASPERA study is a multicenter, observational, both retrospective and prospective real-world study involving acute ischemic stroke patients occurring on oral anticoagulation. The study will encompass a retrospective (ASPERA-R) and prospective (ASPERA-P) data collection. Patient will be recruited consecutively at different emergency services and stroke units worldwide. University of L'Aquila (UnivAQ) will be in charge of study coordination, data analysis and management. The duration of ASPERA-R will be of 5-year from the study initiation of the study. Participating centers will be given a 6-month timeframe to enter retrospective data, commencing from the date of study approval.

ASPERA-P duration will be of 2 years of enrollment from the study approval and follow-up of 5 years. (study conclusion after 7 years of approval). Inclusion criteria will be: 1.Confirmed diagnosis of ischemic stroke. 2. Availability of at least one neuroimaging exam positive for ischemic lesion(s) consistent with patient symptoms. 3. Ongoing oral anticoagulation at the time of the index ischemic stroke. 4. Prior diagnosis of atrial fibrillation or other cardioembolic arrhythmias. 5. Written informed consent provided by the patient himself or by proxy. Patients with Symptoms not indicative of acute stroke, ongoing intravenous or subcutaneous anticoagulation at the time of stroke will be excluded. ASPERA-R: characterization of demographic, clinical and neuroimaging features of ischemic stroke cases occurring on oral anticoagulants. The primary outcome will be: ASPERA-R : characterization of demographic, clinical and neuroimaging features of ischemic stroke cases occurring on oral anticoagulants. ASPERA-P: risk of ischemic stroke recurrence of ischemic stroke cases occurring on oral anticoagulants across different secondary preventive strategies (i.e., maintaining the same type of oral anticoagulation versus switching to a different secondary prevention strategy) at 90 days, 1 and 5 years after the index stroke. Additionally, the study will aim to investigate the risk of safety events (hemorrhagic transformation, intracranial hemorrhage, other major bleeding events, any bleeding events, death due to any cause), risk of other major ischemic events (transient ischemic attack, myocardial infarction, death due to vascular causes) at each follow-up and to identify demographic, clinical and neuroimaging features of ischemic stroke recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of the index ischemic stroke.
* Confirmed diagnosis of ischemic stroke according to the World Health Organization (WHO) definition.
* Availability of at least one neuroimaging exam (either a non-contrast computed tomography [NCCT] or magnetic resonance imaging [MRI] of the brain) demonstrating one or more ischemic lesions consistent with patient symptoms.
* Ongoing oral anticoagulation at the time of the index ischemic stroke, defined as the last intake within 48 hours prior to stroke symptom onset for patients on direct oral anticoagulants (DOACs), or an international normalized ratio (INR) of ≥1.5 in patients on vitamin K antagonists (VKAs), regardless of the time elapsed between the last intake and stroke symptom onset.
* Prior diagnosis of AF or other cardioembolic arrhythmias.

Exclusion Criteria:

* Symptoms not indicative of acute stroke (i.e., syncope, tonic or clonic activity, dizziness alone, confusion and amnesia alone, chronic or subacute development of focal neurological deficit).
* Ongoing parenteral (intravenous or subcutaneous) anticoagulation at the time of the index event, including bridging with heparin in patients initiating VKA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from various recruiting sites worldwide. All consecutive ischemic stroke patients receiving oral anticoagulation therapy for atrial fibrillation or other cardioembolic arrhythmias at the time of the index stroke who meet the inclusion criteria will be eligible, regardless of hospitalization status. The decision to enroll a patient will be made by local investigators, who must ensure that each candidate meets the study's eligibility requirements.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-02-12 (Estimated); Study Completion 2031-02-12 (Estimated)

PRIMARY OUTCOMES:
ASPERA-R Primary Outcome Measure: Baseline demographic characteristics | At the baseline (index ischemic stroke onset/hospital admission)
  Baseline demographic characteristics of ischemic stroke cases occurring on oral anticoagulants: mean age (years), sex (proportion of males and females), ethnicity (proportion of non-Hispanic White, Hispanic White, Black, Asian, other ethnicities), mean weight (Kg), mean height (cm), median BMI
ASPERA-R Primary Outcome Measure: Baseline clinical characteristics | At the baseline (index ischemic stroke onset/hospital admission)
  Baseline clinical characteristics: type of oral anticoagulation at the time of index ischemic stroke (proportion of patients on DOAC or VKA), ischemic stroke clinical severity (median National Insititue of Health Stroke Scale - NIHSS), type of clinical presentation (proportion of patients with anterior or posterior circulation stroke), competing stroke etiology (proportion of patients with large-artery-atherosclerosis or lacunar or other determined or undetermined etiology), risk factors (proportion of patients with hypertension, dyslipidemia, diabetes, history of prior stroke/transient ischemic attack, ischemic cardiopaty, peripheral artery disease, chronic kidney or liver failure), acute ischemic stroke treatment (proportion of patients who undergo intravenous thrombolysis or endovascular thrombectomy)
ASPERA-R Primary Outcome Measure: Baseline Neuroimaging characteristics | At the baseline (index ischemic stroke onset/hospital admission)
  Baseline Neuroimaging characteristics: large vessel occlusion (proportion of patients with large vessel occlusion), site of large vessel occlusion (proportion of patients with anterior or middle or posterior cerebral arteries occlusion), degree of large vessel occlusion (according to the modified treatment in cerebral infarction - mTICI - score: from 0 - no perfusion - to 3 - complete perfusion), median number of new ischemic lesion(s) at neuroimaging, site of new ischemic lesion(s) at neuroimaging (anterior or posterior circulation, right or left hemisphere or bilateral), presence of hemorrhagic infarction at neuroimaging, degree of hemorrhagic infarction at neuroimaging (according to the Heidelberg classification system: Hemorrhagic Infarction - Small petechiae along the margins of the infarcted area or more confluent petechiae without space-occupying effect (HI2). Parenchymal Hematoma - A hematoma covering less (PH1) or more (PH2) than 30% of the infarcted area.
ASPERA-P Primary Outcome Measure: New ischemic stroke or transient ischemic attack | 90-day, 1-year and 5-year post-stroke
  New ischemic stroke or transient ischemic attack (proportion of patients with new ischemic stroke or transient ischemic attack)

SECONDARY OUTCOMES:
ASPERA-R Secondary Outcome Measure: All-cause mortality | Discharge and 90-day post-stroke
  All-cause mortality (proportion of patients who died due to any cause)
ASPERA-R Secondary Outcome Measure: Vascular death | Discharge and 90-day post-stroke
  Vascular death (death due to stroke, myocardial infarction, pulmonary embolism, sudden death or arrhythmias)
ASPERA-R Secondary Outcome Measure: New ischemic stroke or transient ischemic attack | Discharge and 90-day post-stroke
  New ischemic stroke or transient ischemic attack (proportion of patients with new ischemic stroke or transient ischemic attack)
ASPERA-R Secondary Outcome Measure: Myocardial infarction | Discharge and 90-day post-stroke
  Myocardial infarction (proportion of patients with any type of myocardial infarction)
ASPERA-R Secondary Outcome Measure: Moderate-to-severe bleeding events | Discharge and 90-day post-stroke
  Moderate-to-severe bleeding events (proportion of patients with moderate-to-severe bleedings as defined according to the GUSTO bleeding classification): GUSTO severe or life-threatening bleeding is defined as either intracranial haemorrhage or bleeding resulting in haemodynamic compromise necessitating intervention. GUSTO moderate bleeding is defined as bleeding requiring transfusion, but not resulting in haemodynamic compromise.
ASPERA-R Secondary Outcome Measure: Intracranial hemorrhage | Discharge and 90-day post-stroke
  Intracranial hemorrhage (any type of intracranial hemorrhage)
ASPERA-R Secondary Outcome Measure: Ordinal distribution of modified Rankin Scale scores | Discharge and 90-day post-stroke
  Ordinal distribution of modified Rankin Scale scores (proportion of patients within each category of the modified Rankin Scale): Symptoms without any disability (score of 1), Symptoms with mild disability (score of 2), Symptoms with mild-to-moderate disability (score of 3), Symptoms with moderate-to-severe disability (score of 4), Symptoms with severe disability (score of 5), Death (score of 6)
ASPERA-P Secondary Outcome Measure: All-cause mortality | 90-day, 1-year and 5-year post-stroke
  All-cause mortality (proportion of patients who died due to any cause)
ASPERA-P Secondary Outcome Measure: Vascular death | 90-day, 1-year and 5-year post-stroke
  Vascular death (death due to stroke, myocardial infarction, pulmonary embolism, sudden death or arrhythmias)
ASPERA-P Secondary Outcome Measure: Myocardial infarction | 90-day, 1-year and 5-year post-stroke
  Myocardial infarction (proportion of patients with any type of myocardial infarction)
ASPERA-P Secondary Outcome Measure: Intracranial Hemorrhage | 90-day, 1-year and 5-year post-stroke
  Intracranial hemorrhage (any type of intracranial hemorrhage)
ASPERA-P Secondary Outcome Measure: Moderate-to-severe bleeding events | 90-day, 1-year and 5-year post-stroke
  Moderate-to-severe bleeding events (proportion of patients with moderate-to-severe bleedings as defined according to the GUSTO bleeding classification): GUSTO severe or life-threatening bleeding is defined as either intracranial haemorrhage or bleeding resulting in haemodynamic compromise necessitating intervention. GUSTO moderate bleeding is defined as bleeding requiring transfusion, but not resulting in haemodynamic compromise.
ASPERA-P Secondary Outcome Measure: Minor bleeding events | 90-day, 1-year and 5-year post-stroke
  Minor bleeding events (proportion of patients with minor bleedings as defined according to the GUSTO bleeding classification): Any bleedings that is not intracranial haemorrhage or bleeding resulting in haemodynamic compromise necessitating intervention, or bleeding requiring transfusion.
ASPERA-P Secondary Outcome Measure: Any bleeding events | 90-day, 1-year and 5-year post-stroke
  Any bleeding events (proportion of patients with any bleedings irrespective of their severity)
ASPERA-P Secondary Outcome Measure: Ordinal modified Rankin Scale scores distribution | 90-day, 1-year and 5-year post-stroke
  Ordinal distribution of modified Rankin Scale scores (proportion of patients within each category of the modified Rankin Scale): Symptoms without any disability (score of 1), Symptoms with mild disability (score of 2), Symptoms with mild-to-moderate disability (score of 3), Symptoms with moderate-to-severe disability (score of 4), Symptoms with severe disability (score of 5), Death (score of 6)

CONTACTS AND LOCATIONS:
Locations (47):
- Department of Neurology, Sveti Duh University Hospital, Zagreb, Croatia
- Copenhagen University Hospital, Bispebjerg Hospital, Copenhagen, Denmark
- Egypt (3):
  - Neurology Department, Assiut University Hospitals, Asyut
  - Neurology Department, Faculty of Medicine , Ain Shams University, Cairo
  - Neurology Unit, Kobry Elkoba Medical Complex, Cairo
- Université Cote d'Azur UR2CA-URRIS, Unité Neurovasculaire, CHU Hôpital Pasteur 2, Nice, France
- Germany (2):
  - Department of Neurology, Charite, Berlin Germany and Center for Stroke Research (CSB), Berlin
  - Department of Neurology, Martin-Luther-University of Halle-Wittenberg, Halle
- Italy (24):
  - Neurological Clinic, Marche Polytechnic University, Ancona
  - SC Neurologia, Stroke Unit, Ospedale di Venere, Bari
  - IRCCS Istituto delle Scienze Neurologiche, Bologna
  - SCA Neurologia, USL Umbria 1, Città di Castello
  - Azienda Ospedaliero-Universitaria di Ferrara, Arcispedale Sant'Anna, Ferrara
  - SOD Stroke Unit, Azienda Ospedaliero Universitaria Careggi, Florence
  - Stroke Unit, Hospital Fabrizio Spazian, Frosinone
  - University of L'Aquila, L’Aquila
  - Neurology and Stroke Unit, ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Neurology and Stroke Unit, AORN Antonio Cardarelli, Naples
  - UOC Neurologia e Stroke Unit, AOOR. Villa Sofia - Cervello, Palermo
  - Department of Medicine and Surgery, University of Parma, Parma
  - Department of Emergency Neurology and Stroke Unit, IRCCS C. Mondino, Pavia
  - Medicina Interna e d'Urgenza - Stroke Unit, Azienda Ospedaliera di Perugia, Perugia
  - Department of Emergency Neurology and Stroke Unit, Pescara Hospital, Pescara
  - Department of Neuroscience, Neurology Unit, S.Maria delle Croci Hospital, AUSL Romagna, Ravenna
  - Neurology Unit, Stroke Unit, Azienda Unità Sanitaria Locale-IRCCS di Reggio Emilia, Reggio Emilia
  - UOSD Stroke Unit, Azienda Ospedaliera San Camillo Forlanini, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome
  - UOC Neurologia, Ospedale Provinciale "Madonna del Soccorso", San Benedetto del Tronto
  - UOC Stroke Unit, Emergency and Urgency Department, AOU Senese, Siena
  - ASL Abruzzo 4, G.Mazzini Hospital, Teramo
  - SOSD Stroke Unit, Department of Head, Neck, and Neuroscience, Udine University Hospital, Udine
  - Stroke Unit, Neurologia A, Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- University Clinic of Neurology, University "Ss.Cyril and Methodius"-Faculty of Medicine, Skopje, North Macedonia
- Department of Neurology, Jagiellonian University Medical College, Krakow, Poland
- Portugal (2):
  - Lisbon Central University Hospital - ULS São José and Faculdade de Medicina, Universidade de Lisboa, Lisbon
  - Hospital de Santa Maria, Lisbon
- Elias University Emergency Hospital, Carol Davila University of Medicine and Pharmacy, Bucharest, Romania
- Saudi Arabia (2):
  - King Abdulaziz Medical City, Riyadh
  - Vascular Neurology Division National Neuroscience Institute King Fahad Medical City, Riyadh
- Department of Neurology, Faculty of Medicine, P. J. Safarik University and University Hospital L. Pasteur, Košice, Slovakia
- Spain (2):
  - La Paz University Hospital, Universidad Autónoma de Madrid, IdiPAZ Research Institute, Madrid
  - Department of Medicine, University of Valladolid, Valladolid
- University Teaching Hospital St. Gallen, Sankt Gallen, Switzerland
- United Kingdom (4):
  - Southmead Hospital, North Bristol NHS Trust, Bristol, UK
  - St George's University Hospitals NHS Foundation Trust, London, UK
  - Department of Brain Sciences, Imperial College London, London, UK
  - Department of Stroke and Neuroscience, Charing Cross Hospital, Imperial College, London, UK

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual clinical data collected in the study with other researchers upon reasonable request, in line with ethical guidelines and data protection regulations. Data will be de-identified to protect participant confidentiality.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: From the end of the ASPERA-P study (10/02/2029) up to 10 years (10/02/2039)
Access Criteria: Access will be granted for purposes of replicating findings, conducting meta-analyses, or pursuing related research questions, subject to approval by the study's data governance committee and appropriate institutional review boards. Researchers will be required to sign data-sharing agreements to ensure proper use and compliance with confidentiality standards.